CLINICAL TRIAL: NCT00191555
Title: Double-Blind Long-term Study Comparing the Efficacy and Safety of Olanzapine Versus Haloperidol in Patients With Schizophrenia Previously Stabilized With Conventional Antipsychotic Treatment
Brief Title: Efficacy Study of Switching Stabilized Schizophrenic Patients From Conventional to Atypical Antipsychotic Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6589; F1D-FP-S029
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2006-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine; Haloperidol

INTERVENTIONS:
Drug: olanzapine
Drug: haloperidol

SUMMARY:
The objective of this study is to demonstrate that there is a benefit in switching chronic schizophrenic patients from conventional antipsychotic to olanzapine in terms of efficacy, neurological safety and patient's outcome.

ELIGIBILITY:
Inclusion Criteria:

Schizophrenic patient meeting the DSM-IV diagnostic criteria more than one year ago and treated with antipsychotic for at least 1 year.

Outpatient (or patient admitted to hospital for social or logistic reasons).

Patient receiving a stable dose of the same conventional antipsychotic for at least 8 weeks before visit 1.

Patient presenting a PANSS score equal or greater than 49 at Visit 2.

Patient considered by the investigator as possible candidates for a switch, owing to inadequate efficacy or poor safety of the current treatment.

Exclusion Criteria:

Patient presenting a schizophreniform or a schizo-affective disorder according to the DSM-IV diagnostic criteria, or any other disorder from Axis I of the DSM-IV, or a disorder from Axis II (limit personality), substance dependence or substance abuse.

Administration of an atypical antipsychotic drug during the 8 weeks preceding V1.

History of resistance to antipsychotic drugs

Hospitalization in a psychiatric unit or in a psychiatric emergency department within the 8 weeks preceding the beginning of the study.

Presence of serious unstable disease, such as a fatal outcome or hospitalization in an intensive care unit, is foreseeable within a period of 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360
Dates: Start 2003-08; Study Completion 2006-05

PRIMARY OUTCOMES:
The primary efficacy measure is defined as relapse. Relapse is defined by the presence of at least one of the following criteria:
Psychiatric hospitalization.
A 25% increase in the total score on the PANSS scale (Kay SR et al. 1987) in relation to the score obtained at the baseline visit (Visit 2).
A major deterioration in clinical condition, defined by a score of 6 ("much worse") or 7 ("very much worse") on the CGI-I scale (Clinical Global Impression-Improvement)
Suicide attempt requiring medical treatment and/or jeopardizing vital prognosis (self-mutilation, ingestion of a toxic substance, defenestration, self-mutilation with suicidal intent).

SECONDARY OUTCOMES:
The following secondary efficacy criteria will be measured at the times indicated in the Schedule of Events
Positive and negative symptom scale : PANSS
Clinical global impression scale: CGI [Clinical global impression-severity of illness (CGI-S); Clinical global impression-improvement of illness (CGI-I); Clinical Global Impression scale - Psychic distress]
Schizophrenic Communication Disorder Rating Scale: SCD
Social Interactions measurement tools
Intention Reading Task in a real-life situation
Patient Outcome based on Preference Tool: POP
Patient's quality of life: S-QOL

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (62):
- France (62):
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Aix-en-Provence
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Alençon
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Alise-Sainte-Reine
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Amilly
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Aubergenville
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Barbazan-Debat
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Bohars
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Bordeaux
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Bourges
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Bron
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Brumath
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Castres
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Challans
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Chaumont
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Château-Gontier
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Cluses
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Decize
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Dijon
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Dole
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Figeac
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Fontaines
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Graulhet
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Hénin-Beaumont
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, L'Aigle
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, La Roche-sur-Foron
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, La Rochelle
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, La Seyne-sur-Mer
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Limoges
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Longuic
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Mably
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Marseille
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Melun
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Metz
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Mont-Saint-Martin
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Montéléger
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Montfavet
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Montpellier
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Mulhouse
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Nancy
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Narbonne
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Nevers
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Niort
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Paris
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Plaisir
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Poitiers
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Pont-à-Mousson
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Reims
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Saint-Cyr-au-Mont-d'Or
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Saint-Égrève
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Saint-Julien-en-Genevois
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Saint-Nazaire
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Sète
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Sin-le-Noble
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, St-Malo
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Strasbourg
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Tarbes
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Torcy
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Toulon
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Toulouse
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Vaulx-en-Velin
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Viersat
  - Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Villejuif

REFERENCES:
- [Derived] Ibragimov K, Keane GP, Carreno Glaria C, Cheng J, Llosa AE. Haloperidol (oral) versus olanzapine (oral) for people with schizophrenia and schizophrenia-spectrum disorders. Cochrane Database Syst Rev. 2024 Jul 3;7(7):CD013425. doi: 10.1002/14651858.CD013425.pub2. PMID 38958149